CLINICAL TRIAL: NCT03575364
Title: ClotTriever Outcomes (CLOUT) Registry
Acronym: CLOUT
Status: Completed | Type: Observational
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-001
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Deep Vein Thrombosis Leg; DVT; Chronic DVT of Lower Extremity; Acute DVT of Lower Extremity
Keywords: ClotTriever; Thrombectomy
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Analysis Population: Patients with unilateral acute or subacute DVT of less than or equal to 6 weeks' duration without recent (≤ 3 month) history of venous intervention.
  Interventions: Device: ClotTriever
- Full Analysis Population: Subjects with proximal lower extremity DVT involving the femoral, common, femoral, iliac veins or inferior vena cava (IVC), alone or in combination.
  Interventions: Device: ClotTriever

INTERVENTIONS:
Device: ClotTriever — Thrombectomy

SUMMARY:
Evaluate real world patient outcomes after treatment of acute, subacute, and chronic proximal lower extremity deep vein thrombosis (DVT) with the ClotTriever Thrombectomy System.

DETAILED DESCRIPTION:
The CLOUT Registry is a prospective, multi-center, observational registry of subjects with proximal lower extremity DVT treated with the ClotTriever Thrombectomy System. The Registry will collect data on demographics, comorbidities, details from the DVT diagnosis and treatment, and clinical outcomes through 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Proximal lower extremity DVT involving the femoral, common femoral, iliac veins, or inferior vena cava (IVC), alone or in combination.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Prior venous stent in the target venous segment
* IVC aplasia/hypoplasia or other congenital anatomic anomalies of the IVC or iliac veins
* IVC filter in place at the time of the planned index procedure
* Allergy, hypersensitivity, or thrombocytopenia from heparin or iodinated contrast agents, except for mild to moderate contrast allergies for which pretreatment can be used
* Life expectancy less than 1 year
* Chronic non-ambulatory status
* Known hypercoagulable states that, in the opinion of the Investigator, cannot be medically-managed throughout the study period
* Unavailability of a lower extremity venous access site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proximal lower extremity DVT.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Dexter, MD, Principal Investigator — Sentara Vascular Specialists; Robert Beasley, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (43):
- United States (43):
  - St. Vincent's East, Birmingham, Alabama
  - Affinity Cardiovascular Specialists, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - Vascular and Interventional Specialists of Orange County, Orange, California
  - University of Colorado, Denver, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - MedStar Health Research Institution, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Lakeland Vascular Institute, Lakeland, Florida
  - Mount Sinai Medical Center of Florida, Miami Beach, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Longstreet Clinic, Gainesville, Georgia
  - Wesley Medical Center, Wichita, Kansas
  - Surgical Care Associates, Louisville, Kentucky
  - Lafayette General, Lafayette, Louisiana
  - Opelousas General, Opelousas, Louisiana
  - McLaren Bay Heart and Vascular, Bay City, Michigan
  - Millenium Cardiology, Farmington Hills, Michigan
  - Ascension Genesys Hospital, Grand Blanc, Michigan
  - Beaumont Health, Royal Oak, Michigan
  - University of Missouri, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Lee's Summit, Missouri
  - Washington University at St. Louis, St Louis, Missouri
  - Hackensack Meridian, Hackensack, New Jersey
  - Albany Medical College, Albany, New York
  - SUNY, The University at Buffalo, Buffalo, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Northwell Health, Staten Island, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Mercy Health - The Heart Institute, Fairfield, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Thomas Jefferson, Philadelphia, Pennsylvania
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - Methodist Healthcare Foundation, Germantown, Tennessee
  - Houston Healthcare Medical Center, Houston, Texas
  - University of Texas Health Sciences Center - Houston, Houston, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Providence Sacred Heart, Spokane, Washington
  - Gunderson Health, La Crosse, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dexter DJ, Kado H, Schor J, Annambhotla S, Olivieri B, Mojibian H, Maldonado TS, Gandhi S, Paulisin J, Bunte MC, Angel W, Roberts J, Veerina K, Abramowitz S, Elmasri F, Hnath J, Jung M, Long D, Sanchez L, Cosme O, Skripochnik E, Lodha A, Shaikh A, King C, Bisharat M, Beasley RE; CLOUT Investigators. Interim outcomes of mechanical thrombectomy for deep vein thrombosis from the All-Comer CLOUT Registry. J Vasc Surg Venous Lymphat Disord. 2022 Jul;10(4):832-840.e2. doi: 10.1016/j.jvsv.2022.02.013. Epub 2022 Feb 24. PMID 35218955
- [Background] Maldonado TS, Dexter DJ, Kado H, Schor J, Annambhotla S, Mojibian H, Beasley RE; CLOUT Registry Investigators. Outcomes from the ClotTriever Outcomes Registry show symptom duration may underestimate deep vein thrombus chronicity. J Vasc Surg Venous Lymphat Disord. 2022 Nov;10(6):1251-1259. doi: 10.1016/j.jvsv.2022.04.015. Epub 2022 Jun 14. PMID 35714903
- [Background] Dexter D, Kado H, Shaikh A, Schor J, Annambhotla S, Zybulewski A, Paulisin J, Bisharat M, Mouawad NJ, Bunte MC, Maldonado T, Skripochnik E, Raskin A, Gandhi S, Ichinose E, Beasley R, Mojibian H. Safety and Effectiveness of Mechanical Thrombectomy From the Fully Enrolled Multicenter, Prospective CLOUT Registry. J Soc Cardiovasc Angiogr Interv. 2023 Feb 23;2(2):100585. doi: 10.1016/j.jscai.2023.100585. eCollection 2023 Mar-Apr. PMID 39129803
- [Background] Abramowitz SD, Kado H, Schor J, Annambhotla S, Mojibian H, Marino AG, Maldonado TS, Gandhi S, Paulisin J, Bunte MC, Angel W, Roberts J, Veerina K, Long D, Elmasri F, Shaikh A, Beasley RE, Dexter D; CLOUT Investigators. Six-Month Deep Vein Thrombosis Outcomes by Chronicity: Analysis of the Real-World ClotTriever Outcomes Registry. J Vasc Interv Radiol. 2023 May;34(5):879-887.e4. doi: 10.1016/j.jvir.2022.12.480. PMID 37105663
- [Background] Shaikh A, Zybulewski A, Paulisin J, Bisharat M, Mouawad NJ, Raskin A, Ichinose E, Abramowitz S, Lindquist J, Azene E, Shah N, Nguyen J, Cockrell J, Khalsa B, Khetarpaul V, Murrey DA Jr, Veerina K, Skripochnik E, Maldonado TS, Bunte MC, Annambhotla S, Schor J, Kado H, Mojibian H, Dexter D; CLOUT Investigators. Six-Month Outcomes of Mechanical Thrombectomy for Treating Deep Vein Thrombosis: Analysis from the 500-Patient CLOUT Registry. Cardiovasc Intervent Radiol. 2023 Nov;46(11):1571-1580. doi: 10.1007/s00270-023-03509-8. Epub 2023 Aug 14. PMID 37580422
- [Background] Abramowitz S, Marko X, Willis VC, Mills C, Black SA. Association Between 30 Day Villalta Scores and Long Term Post-Thrombotic Syndrome Incidence and Severity Following Acute Deep Vein Thrombosis. Eur J Vasc Endovasc Surg. 2024 Jan;67(1):167-168. doi: 10.1016/j.ejvs.2023.09.045. Epub 2023 Oct 5. No abstract available. PMID 37802419
- [Background] Bisharat MB, Ichinose EJ, Veerina KK, Khetarpaul V, Azene EM, Plotnik AN, Hnath J, Trestman E, Harlin SA, Bhat A, Li S, Long GW, O'Connor D, Winokur RS, Zia S, Dexter DJ. One-Year Clinical Outcomes Following Mechanical Thrombectomy for Deep Vein Thrombosis: A CLOUT Registry Analysis. J Soc Cardiovasc Angiogr Interv. 2024 Feb 15;3(3Part A):101307. doi: 10.1016/j.jscai.2024.101307. eCollection 2024 Mar. PMID 39131784
- [Background] Abramowitz S, Bunte MC, Maldonado TS, Skripochnik E, Gandhi S, Mouawad NJ, Mojibian H, Schor J, Dexter DJ; CLOUT study collaborators. Mechanical Thrombectomy vs. Pharmacomechanical Catheter Directed Thrombolysis for the Treatment of Iliofemoral Deep Vein Thrombosis: A Propensity Score Matched Exploratory Analysis of 12 Month Clinical Outcomes. Eur J Vasc Endovasc Surg. 2024 Apr;67(4):644-652. doi: 10.1016/j.ejvs.2023.11.017. Epub 2023 Nov 21. PMID 37981003
- [Background] Abramowitz S, Shaikh A, Mojibian H, Mouawad NJ, Bunte MC, Skripochnik E, Lindquist J, Elmasri F, Khalsa B, Bhat A, Nguyen J, Shah N, Noor SS, Murrey D, Gandhi S, Raskin A, Schor J, Dexter DJ. Comparison of anticoagulation vs mechanical thrombectomy for the treatment of iliofemoral deep vein thrombosis. J Vasc Surg Venous Lymphat Disord. 2024 Jul;12(4):101825. doi: 10.1016/j.jvsv.2024.101825. Epub 2024 Jan 24. PMID 38278173
- See also: Six-Month Deep Vein Thrombosis Outcomes by Chronicity: Analysis of the Real-World ClotTriever Outcomes Registry. — http://doi.org/10.1016/j.jvir.2022.12.480
- See also: Safety and Effectiveness of Mechanical Thrombectomy From the Fully Enrolled Multicenter, Prospective CLOUT Registry. — https://doi.org/10.1016/j.jscai.2023.100585
- See also: Interim outcomes of mechanical thrombectomy for deep vein thrombosis from the All-Comer CLOUT Registry. — https://doi.org/10.1016/j.jvsv.2022.02.013
- See also: Outcomes from the ClotTriever Outcomes Registry show symptom duration may underestimate deep vein thrombus chronicity. — https://doi.org/10.1016/j.jvsv.2022.04.015
- See also: Six-Month Outcomes of Mechanical Thrombectomy for Treating Deep Vein Thrombosis: Analysis from the 500-Patient CLOUT Registry. — http://doi.org/10.1007/s00270-023-03509-8
- See also: Mechanical Thrombectomy vs. Pharmacomechanical Catheter Directed Thrombolysis for the Treatment of Iliofemoral Deep Vein Thrombosis: A Propensity Score Matched Exploratory Analysis of 12 Month Clinical Outcomes — https://doi.org/10.1016/j.ejvs.2023.09.045
- See also: Association Between 30 Day Villalta Scores and Long Term Post-Thrombotic Syndrome Incidence and Severity Following Acute Deep Vein Thrombosis — https://doi.org/10.1016/j.ejvs.2023.09.045
- See also: Comparison of anticoagulation vs mechanical thrombectomy for the treatment of iliofemoral deep vein thrombosis. — https://pubmed.ncbi.nlm.nih.gov/38278173/
- See also: One-Year Clinical Outcomes Following Mechanical Thrombectomy for Deep Vein Thrombosis: A CLOUT Registry Analysis — https://doi.org/10.1016/j.jscai.2024.101307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients presenting to the hospital/emergency department with proximal lower extremity deep vein thrombosis (DVT) and meeting all eligibility requirements for enrollment in the CLOUT study.
Pre-assignment Details: The first 91 subjects with unilateral acute or subacute DVT of less than or equal to 6 weeks' duration without recent (≤ 3 month) history of venous intervention were enrolled in the Primary Analysis Population. Once the Primary Analysis Population was fully accrued, subjects meeting the study criteria continued to be enrolled and were evaluated as part of the Full Analysis Population.
Groups:
- Full Analysis Population: The Full Analysis Population consists of 499 subjects with proximal lower extremity DVT involving the femoral, common femoral, iliac veins or inferior vena cava (IVC), alone or in combination.
Period: Overall Study
Arm/Group | Full Analysis Population
Started | 499
Primary Analysis Population (The Primary Analysis Population is a subset of the Full Analysis Population, comprising the first 91 subjects with unilateral acute or subacute DVT of less than or equal to 6 weeks duration without recent (≤ 3 month) history of venous intervention.) | 91
Primary Safety Cohort (The Primary Safety Cohort are the 76 subjects in the Primary Analysis Population who had evaluable data for the primary safety endpoint.) | 76
Primary Effectiveness Cohort (The Primary Effectiveness Cohort are the 89 subjects in the Primary Analysis Population with core laboratory-documented intraluminal thrombus at pre- and post- index procedure who have at least one target venous segment (TVS) treated with the study device.) | 89
Full Analysis Population (The Full Analysis Population consists of 499 subjects with proximal lower extremity DVT involving the femoral, common femoral, iliac veins or inferior vena cava (IVC), alone or in combination.) | 499
Completed | 285
Not Completed | 214
Not completed — Death | 45
Not completed — Lost to Follow-up | 114
Not completed — Withdrawal by Subject | 21
Not completed — Physician Decision | 11
Not completed — Subject Refused Follow-up | 13
Not completed — Hospital Administration decision, Research department closed | 6
Not completed — Patient moved out of the state | 1
Not completed — Patient no longer has insurance, will not return to clinic. | 1
Not completed — Patient is lost to follow up | 1
Not completed — Patient was unable to get to the clinic due to health problems and transportation difficulties | 1

BASELINE CHARACTERISTICS:
Arm/Group | Full Analysis Population
Number analyzed (Participants) | 499
Age, Continuous [Median (Full Range); unit: years] | 61.85 [18.6 to 98.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252
  Male | 247
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska | 4
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 101
  White | 374
  More than one race | 2
  Other | 4
  Unknown or Missing | 11
Height (cm) [Median (Full Range); unit: cm] — Population: Fewer participants were analyzed due to missing baseline height data.
  cm
    number analyzed (Participants) | 492
    (all) | 170.20 [147.3 to 200.7]
Weight (kg) [Median (Full Range); unit: kg] — Population: Fewer participants were analyzed due to missing baseline weight data.
  kg
    number analyzed (Participants) | 498
    (all) | 88.50 [44.8 to 178.5]
BMI (kg/m^2) [Median (Full Range); unit: kg/m^2] — Population: Baseline BMI data were missing for 7 subjects .
  kg/m^2
    number analyzed (Participants) | 492
    (all) | 30.203 [17.24 to 62.35]

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Proportion Participants With Major Adverse Events
Description: The primary safety endpoint is the proportion of participants with Major Adverse Events (MAE). MAEs are defined as a composite endpoint triggered when any of four categories of events occurred through 30 days after the index procedure, as observed in the Primary Safety Cohort (the composite endpoints were not observed for the Full Analysis Population:
  * All-cause mortality
  * Major bleeding
  * New symptomatic pulmonary embolism (PE) documented by computed tomography pulmonary angiography (CTPA)
  * Rethrombosis of a target vessel segment (TVS)
Time Frame: 30 days
Population: The Primary Analysis Population is a subset of the Full Analysis Population, comprising the first 91 subjects with unilateral acute or subacute DVT of less than or equal to 6 weeks duration without recent (≤ 3 month) history of venous intervention.
  The Primary Safety Cohort are the 76 subjects in the Primary Analysis Population who had evaluable data for the primary safety endpoint.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Safety Cohort: Subjects from the Primary Analysis Population who had evaluable data for the primary safety endpoint.
Arm/Group | Primary Safety Cohort
Number analyzed (Participants) | 76
Participants | 15

2. Secondary Outcome: Primary Effectiveness Endpoint (Primary Effectiveness Cohort): Participants With Complete or Near Complete (≥75%) Removal of Venous Thrombus
Description: Complete or near complete (≥75%) removal of venous thrombus from the TVS, as determined by the percent reduction in the Marder score for those segments. When more than one venous segment is treated, the change in Marder score is calculated as the total score for the treated segments prior to intervention with the study device (baseline score) minus the total score after treatment with the study device but before treatment with any adjunctive devices or pharmacologic agents (post-treatment score), divided by the baseline score.
Time Frame: Index Procedure (approximately 0.5 hours on day 0)
Population: The Primary Analysis Population is a subset of the Full Analysis Population is the first 91 subjects with unilateral acute or subacute DVT of less than or equal to 6 weeks duration without recent (≤ 3 months) history of venous intervention.
  The Primary Effectiveness Cohort are the 89 subjects in the Primary Analysis Population with core laboratory-documented intraluminal thrombus at pre- and post- index procedure who have at least one target venous segment (TVS) treated with the study device.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Effectiveness Cohort: Subjects from the Primary Analysis Population with core laboratory-documented intraluminal thrombus at pre- and post- index procedure who have at least one target venous segment (TVS) treated with the study device.
Arm/Group | Primary Effectiveness Cohort
Number analyzed (Participants) | 89
Participants | 68

3. Other Pre Specified Outcome: Primary Effectiveness Endpoint (Full Analysis Population): Participants With Complete or Near Complete (≥75%) Removal of Venous Thrombus
Description: as for outcome 2
Time Frame: Index Procedure (approximately 0.5 hours on day 0)
Population: The Full Analysis Population consists of 499 subjects with proximal lower extremity DVT involving the femoral, common femoral, iliac veins or inferior vena cava (IVC), alone or in combination.
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Population: Subjects from the Full Analysis Population with evaluable data for the Primary Effectiveness Endpoint (core laboratory-documented intraluminal thrombus at pre- and post- index procedure for at least one TVS treated with the study device). Thirteen (13) subjects did not have evaluable data for this endpoint, yielding 486 analyzed subjects.
Arm/Group | Full Analysis Population
Number analyzed (Participants) | 486
Participants | 443

ADVERSE EVENTS:
Time Frame: All adverse events were assessed at the index procedure, discharge, 30-day, 6-month, 1-year, and 2-year follow-up visits, study exit (regardless of 2-year follow-up visit completion), and any unscheduled visits prior to the 2-year follow-up visit.
Description: This study captured AEs related to the subject's DVT and its treatment. AEs include all events in the primary safety endpoint, all device/procedure-related AEs, and death. AE counts reflect those at study exit.
  Note: 169 patients had unknown mortality status due to withdrawal or loss to follow-up before completing all study visits. The all-cause mortality rate at study exit among patients with confirmed mortality status was 13.6% (45/330).
Arm/Group | Full Analysis Population
All-Cause Mortality (participants affected / at risk) | 45/330
Serious Adverse Events (participants affected / at risk) | 120/499
Other Adverse Events (participants affected / at risk) | 76/499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Analysis Population (N=499)
Deep vein thrombosis (Vascular disorders) | 68 (68)
Pulmonary embolism (Vascular disorders) | 11 (11)
Cerebrovascular accident (Vascular disorders) | 3 (3)
Blood loss anaemia (Vascular disorders) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1)
Extrinsic iliac vein compression (Vascular disorders) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 1 (1)
Spontaneous haematoma (Vascular disorders) | 1 (1)
Vascular stent occlusion (Vascular disorders) | 1 (1)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Malignant neoplasm of pleura metastatic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Death (General disorders) | 7 (7)
Vascular stent stenosis (General disorders) | 1 (1)
Septic shock (Infections and infestations) | 3 (3)
Meningitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Spinal cord infection (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Pancreatic carcinoma (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Analysis Population (N=499)
Deep vein thrombosis (Vascular disorders) | 76 (76)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03575364/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT03575364/SAP_001.pdf